CLINICAL TRIAL: NCT04574128
Title: Blood Loss With Cardiopulmonary Bypass, Re-transfusion or Not.
Brief Title: Retransfusion or Not of Cardiotomy Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ECC 2020
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Intervention Model Description: Randomised controlled non-inferiority trial
Who Masked: Participant, Care Provider
Masking Description: The person that controle the heart- and lung mashine is not masked. Other members of the surgical team is masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retransfusion of cardiotomy blood or not (Experimental): Intervention group does not get cardiotomy blood retransfusion via heart-and lung machine while control does.
  Interventions: Procedure: No retransfusion of cardiotomy blood
- No retransfusion of cardiotomy blood (No Intervention)

INTERVENTIONS:
Procedure: No retransfusion of cardiotomy blood — No retransfusion of cardiotomy blood via heart- and lung mashine
  Arms: Retransfusion of cardiotomy blood or not

SUMMARY:
This randomised controlled trial has a non-inferiority design. The aim is to test if the blood loss (volume in mL and hemoglobin) is effected by heart and lung cardiotomy retransfusion, or not? Forty CABG (Coronary Artery By pass Grafting) patients will be allocated to either receive retransfusion (n=20) of cardiotomy blood via the heart and lung mashine, or no retransfusion (n=20).

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG.

Exclusion Criteria:

* Anaemia, infection, massive bleeding, CABG off pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
blood loss | During 5 days hemoglobin will be measured as the clinical rutine or as needed.
  Hemoglobin
Blood loss | During 2 days or while surgical drains remains, blood volume in mL is measured.
  Blood volume in millilitre (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Wistrand, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- University Hospital in Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due to ethical considerations of the participant integrity. Bacterial growth can be seen as sensitive data. The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.